CLINICAL TRIAL: NCT06888700
Title: Project on tDCS Intervention to Enhance Advanced Social Cognitive Functions in Drug Rehabilitation Individuals
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Shaanxi Normal University (Other)
Collaborators: Nanyang Technological University (Other)
Responsible Party: Principal Investigator, Yifan Wang, Laboratory Manager, Shaanxi Normal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: L20240186; SFBJYJZXM2023-21-06 (Other Grant/Funding Number: Ministry of Justice in China); 32471114 (Other Grant/Funding Number: The National Natural Science Foundation of China)
Record Dates: First submitted 2025-03-10; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Drug Addiction
Keywords: heroin; advanced social cognitive function
MeSH Terms: conditions — Substance-Related Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active group (Active Comparator): The study was sham-controlled, randomized, and double-blind. Participants with HUD were randomly assigned to either the active or sham groups. The DC-STIMULATOR PLUS (neuroConn, Germany) was used to deliver stimulation via saline-soaked sponge electrodes (25 cm², 5×5 cm, 1.5 mA). The anode was positioned over the rTPJ (P6), with the cathode placed on the left sub-occipital region. The stimulation in the active group lasted for 20 min with a 30-s fade-in and a 30-s fade-out. They received five stimulation sessions within one week, with a minimum interval of 24 hours between each session. The tDCS sensitivity questionnaire was used to assess blinding validity.
  Interventions: Device: Transcranial direct current stimulation
- Sham group (Sham Comparator): The study was sham-controlled, randomized, and double-blind. Participants with HUD were randomly assigned to either the active or sham groups. The DC-STIMULATOR PLUS (neuroConn, Germany) was used to deliver stimulation via saline-soaked sponge electrodes (25 cm², 5×5 cm, 1.5 mA). The anode was positioned over the rTPJ (P6), with the cathode placed on the left sub-occipital region.The stimulation in the sham group was set up as a stimulation cycle of 30s fade-in and 30s fade-out, followed by no current stimulation. They received five stimulation sessions within one week, with a minimum interval of 24 hours between each session. The tDCS sensitivity questionnaire was used to assess blinding validity.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — The participant cohort recruited for this study consists of individuals with substance use disorder (SUD), specifically those addicted to drugs. During the intervention phase, this group will adhere to a strict non-pharmacological intervention protocol, meaning they will not receive any form of pharmacotherapy, neurosurgical intervention, or other neuromodulation-based cognitive interventions, including but not limited to techniques such as transcranial magnetic stimulation (TMS) and transcranial direct current stimulation (tDCS). This design aims to ensure the internal validity of the study results and to exclude potential confounding effects of other interventions on neuroplasticity and cognitive function.

SUMMARY:
This project aims to explore key brain functional and biochemical indicators associated with impaired advanced social cognition through an integrated approach encompassing unconscious control, conscious control, cognitive flexibility, problem-solving, and social interaction domains. By incorporating multimodal measures spanning physiological, neural, cognitive, psychological, and behavioral dimensions, we will develop a comprehensive intervention protocol combining course-based brain stimulation and cognitive training. The study will employ a multi-timepoint, multi-level assessment framework to track the enhancement of higher cognitive functions and brain functional recovery in individuals undergoing drug rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* age between 30 and 60 years;
* fulfilling the diagnostic criteria for severe substance use disorder as specified in the Fifth Edition of the Diagnostic and Statistical Manual of Mental Disorders.
* a history of heroin use exceeding ten years, with a daily average intake of at least 0.1 grams.
* abstinence duration of eight months or less, with a positive result of a urine test before entering the rehabilitation center.
* no history of neuromodulation treatments such as tDCS within the past six months.

Exclusion Criteria:

* a history of alcohol dependence, neurological disorders, or other complex psychiatric conditions.
* the presence of intracranial metallic implants or elevated intracranial pressure.
* a history of epilepsy or recent electroencephalogram evidence of epileptiform activity.
* the use of implanted electronic devices, such as pacemakers;.
* scalp hyperalgesia or a tendency toward bleeding.
* severe cardiac conditions.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-03-19 (Estimated); Primary Completion 2025-04-18 (Estimated); Study Completion 2028-11-17 (Estimated)

PRIMARY OUTCOMES:
Cortical activation from fNIRS | From enrollment to the end of treatment at 1 month
Cortical functional connectivity from fNIRS | From enrollment to the end of treatment at 1 month
Inter-brain neural synchronization from fNIRS hyperscaning | From enrollment to the end of treatment at 1 month
EEG power | From enrollment to the end of treatment at 1 month
EEG microstate | From enrollment to the end of treatment at 1 month
Functional connectivity from EEG | From enrollment to the end of treatment at 1 month
Realistic presented problem task score | From enrollment to the end of treatment at 1 month
  Used to measure problem-solving ability
Score on the Group Realistic Problem Solving task | From enrollment to the end of treatment at 1 month
  Used to measure collaborative problem-solving ability
Score on the joint drawing task | From enrollment to the end of treatment at 1 month
  Used to measure interactive collaboration.
Scores on the pattern game task | From enrollment to the end of treatment at 1 month
  Used to measure social cooperation and competition

SECONDARY OUTCOMES:
Pupil response from eye-tracking | From enrollment to the end of treatment at 1 month
Average fixation duration from eye-traking | From enrollment to the end of treatment at 1 month
Fixation time percentage from eye-traking | From enrollment to the end of treatment at 1 month
Alternative use task (AUT) score | From enrollment to the end of treatment at 1 month
  Used to measure problem-solving ability
Score on the Group Alternative Use Task | From enrollment to the end of treatment at 1 month
  Used to measure collaborative problem solving ability
Cognitive flexibility | From enrollment to the end of treatment at 1 month
  Assessed by Wisconsin Card Quest (WCST).
Cognitive inhibition | From enrollment to the end of treatment at 1 month
  Assessed by stroop task
Mind wandering | From enrollment to the end of treatment at 1 month
  Assessed by interpolation task

CONTACTS AND LOCATIONS:
Locations (1):
- Shaanxi Provincial Chang'an Compulsory Isolation Drug Rehabilitation Center, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No
This study is a government-collaborative project involving sensitive personal information of a vulnerable population, and as such, it is imperative to adhere to strict confidentiality protocols. All data collected will be handled in compliance with ethical guidelines and legal requirements to ensure the protection of participants' privacy.